CLINICAL TRIAL: NCT03322020
Title: Androgen Deprivation Therapy, External Beam Radiotherapy and Stereotactic Radiosurgery Boost for Men With Intermediate- or High-risk Prostate Cancer
Brief Title: Androgen Deprivation Therapy, External Beam Radiotherapy and Stereotactic Radiosurgery Boost for Prostate Cancer
Acronym: ADEBAR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young Seok Kim, Associate professor, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2016-0351-0001
Record Dates: First submitted 2017-10-17; First posted 2017-10-26 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Neoplasm, Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CK 18 Gy (Experimental): Patients who receive Cyberknife boost dose of 18 Gy in 3 fractions
  Interventions: Radiation: Cyberknife boost 18 Gy
- CK 21 Gy (Experimental): Patients who receive Cyberknife boost dose of 21 Gy in 3 fractions
  Interventions: Radiation: Cyberknife boost 21 Gy

INTERVENTIONS:
Radiation: Cyberknife boost 18 Gy — pelvis IMRT dose of 44 Gy/20 fx followed by Cyberknife boost 18 Gy/3 fx
  Arms: CK 18 Gy
Radiation: Cyberknife boost 21 Gy — pelvis IMRT dose of 44 Gy/20 fx followed by Cyberknife boost 21 Gy/3 fx
  Arms: CK 21 Gy

SUMMARY:
For the treatment for intermediate- and high-risk prostate cancer, Cyberknife boost will be used after 4 weeks of intensity modulated radiotherapy to pelvis. The boost doses are 18 Gy and 21 Gy in 3 fractions, respectively. The investigators plan to evaluate the toxicity of two dose groups and decide the appropriate dose for Cyberknife boost. Also, PSA control will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed intermediate- or high-risk prostate cancer within 6 months after enrollment
* ECOG performance status 0-1
* Appropriate values of blood tests within 6 months after enrollment Absolute neutrophil count (ANC) ≥ 1500 cells/mm3 Platelets ≥ 50,000 cells/mm3 Hemoglobin ≥ 8.0 g/dl
* Appropriate values of kidney function within 6 months after enrollment Creatinine < 2.0 ng/dL
* Appropriate values of liver function within 6 months after enrollment total bilirubin < 1.5 X maximum normal value alanine aminotransferase or aspartate aminotransferase < 2.5 X maximum normal value

Exclusion Criteria:

* Presence of distant metastasis
* Presence of pelvic LN metastasis
* History of androgen deprivation therapy within 6 months after enrollment
* History of definitive treatment for prostate cancer (e.g., radical prostatectomy)
* History of pelvic irradiation
* Double primary cancer other than skin/thyroid cancer

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Acute toxicity assessment for 18 Gy and 21 Gy arm | 3 months
  CTCAE v4.03, overactive bladder symptom score (OABSS), International Prostate Symptom Score (IPSS)

SECONDARY OUTCOMES:
Biochemical control free survival | 3 years
  PSA nadir + 2.0ng/ml or Start of salvage hormonal therapy
Late toxicity assessment for 18 Gy and 21 Gy arm | average 6 months
  Late Effects of Normal Tissues (LENT) scoring system

CONTACTS AND LOCATIONS:
Overall Officials: Young Seok Kim, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim YJ, Ahn H, Kim CS, Kim YS. Phase I/IIa trial of androgen deprivation therapy, external beam radiotherapy, and stereotactic body radiotherapy boost for high-risk prostate cancer (ADEBAR). Radiat Oncol. 2020 Oct 8;15(1):234. doi: 10.1186/s13014-020-01665-6. PMID 33032643
- [Derived] Kim YJ, Ahn H, Kim CS, Lee JL, Kim YS. Stereotactic body-radiotherapy boost dose of 18 Gy vs 21 Gy in combination with androgen-deprivation therapy and whole-pelvic radiotherapy for intermediate- or high-risk prostate cancer: a study protocol for a randomized controlled, pilot trial. Trials. 2018 Apr 2;19(1):212. doi: 10.1186/s13063-018-2574-y. PMID 29609646